CLINICAL TRIAL: NCT04640805
Title: Targeted Fortification of Pasteurized Donor Human Milk to Improve Growth in Very Low Birth Weight Infants
Brief Title: Targeted Fortification of Pasteurized Donor Human Milk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/2493
Record Dates: First submitted 2020-11-10; First posted 2020-11-23 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Very Low Birth Weight Infant; Growth Failure; Donor Breast Milk
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Intervention Model Description: Assignment to study group will be done in a 1:1 ratio. Twins/triplets will be randomized to the same group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (standard fortification) (No Intervention): Pasteurized Donor Human Milk (PDHM) will be fortified as per unit protocols, at 1 packet of Human Milk Fortifier (Similac or Pre-Nan) to every 25ml PDHM at a feed volume of 80ml/kg/day
- Intervention group (modified targeted fortification) (Experimental): Pasteurized Donor Human Milk (PDHM) will be analyzed using the Miris Human Milk Analyzer, and PDHM with a fat content of 3.8g/dL or higher will be selected. Additional protein will be added using liquid protein fortifier (Similac) at 1ml to every 25ml PDHM to give an additional 0.67g/dL protein.
  Interventions: Dietary Supplement: Protein supplementation; Other: Analysis with Miris Human Milk Analyzer

INTERVENTIONS:
Dietary Supplement: Protein supplementation — Liquid protein fortifier (Similac) will be added at 1ml per 25ml of PDHM at 130ml/kg/day of feed volume.
  Arms: Intervention group (modified targeted fortification)
Other: Analysis with Miris Human Milk Analyzer — PDHM macronutrient content will be analyzed using the Miris Human Milk Analyzer and PDHM with fat content of 3.8g/dL or higher will be selected and provided.
  Arms: Intervention group (modified targeted fortification)

SUMMARY:
This randomized controlled trial aims to evaluate a modified targeted fortification method of pasteurized donor human milk (PDHM) in very low birth weight infants (VLBWs). Pools of PDHM will be analyzed for macronutrient content using the Miris Human Milk Analyzer. The control arm will receive standard of care, which is PDHM without additional protein fortification. The intervention arm will receive PDHM with a fat content of 3.8g/dL or more, with additional protein fortification of 0.67g/dL. Primary outcome will be rate of malnutrition at hospital discharge or 37 weeks, whichever earlier. Secondary outcomes include body composition, feed tolerance, and morbidity outcomes.

DETAILED DESCRIPTION:
Our hospital milk bank provides pasteurized donor human milk (PDHM) to very low birth weight (VLBW) infants without sufficient mother's milk, with the overall aim of lowering the risk of necrotizing enterocolitis in this population. However, with the introduction of PDHM in our setting, rates of suboptimal weight gain have increased (60.2% to 65.7%). This is likely due to the fact that PDHM is often lower in energy and protein than preterm mother's own milk. One solution to delivery adequate nutrition in this VLBWs receiving PDHM, is targeted fortification, which involves measurement of the macronutrient content of human milk, and adding extra macronutrients to reach nutrient goals. In this proposed study, we will conduct a pilot randomized controlled trial of a modified targeted fortification versus standard care. This study will include preterm VLBW infants (<1500g), without congenital conditions resulting in growth restriction, and receiving >25% of PDHM use in the first week of life. 40 patients in each arm will be recruited over a period of 2 years. The intervention group will receive a modified targeted fortification, consisting of selection of high fat PDHM (3.8g/dL or more) with the addition of protein fortification of 0.67g/dL from week 2 of life until a gestational age of 37 weeks or hospital discharge, whichever earlier. The control group will receive usual regular PDHM with standard fortification using human milk fortifier as per current practice. The primary outcome is the rate of suboptimal growth (drop in weight z-score from birth ≥0.8) at discharge or 37 weeks. Secondary outcomes include body composition, feed tolerance, and morbidity outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight less than or equal to 1500g
* Born at our study hospital or transferred to study hospital within first week of life
* Achieving at least 40ml/kg/day of enteral feeds by day 7 of life
* Receiving at least 25% of pasteurized donor human milk within first 7 days of life

Exclusion Criteria:

* Diagnosed or suspected inborn errors of metabolism
* Acute or chronic renal impairment
* Congenital disease associated with significant growth impairment (including, but not limited to, Trisomy 21, neonatal encephalopathy and seizures, neonatal tumours, achondroplasia, complex congenital heart disease, anorectal malformations, gastrointestinal disorders)

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Malnutrition rate | Hospital discharge or 37 weeks gestation, whichever earlier
  Malnutrition is defined as a decline in weight z-score from birth of 0.8 or more

SECONDARY OUTCOMES:
Linear growth | Hospital discharge or 37 weeks post menstrual age, whichever earlier
  Linear growth will be assessed using z-score changes from birth
Body composition | Hospital discharge or 37 weeks gestation, whichever earlier
  Percent fat mass and fat-free mass measured using air displacement plethysmography
Head circumference growth | Hospital discharge or 37 weeks gestation, whichever earlier
  Head circumference will be assessed using z-score changes from birth
High calorie formula use | Hospital discharge or 35 weeks gestation, whichever earlier
  Proportion of high calorie formula use (e.g. 27kcal/oz or 30kcal/oz formula)
Bronchopulmonary dysplasia | Hospital discharge or 37 weeks gestation, whichever earlier
  Proportion of patients with bronchopulmonary dysplasia
Retinopathy of prematurity | Hospital discharge or 37 weeks gestation, whichever earlier
  Proportion of patients with retinopathy of prematurity

OTHER OUTCOMES:
Neurodevelopmental scores | 18 to 24 months post menstrual age
  Bayley Scales of Infant and Toddler Development scale scores
Infant motor performance | Hospital discharge or 37 weeks gestation, whichever earlier
  Test of Infant Motor Performance scores measured by trained physiotherapists
Duration of hospital stay | Hospital discharge, assessed up to 180 days post menstrual age
  Days of hospital stay, up to 180 days post menstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Chengsi Ong, Principal Investigator — KK Women's and Children's Hospital, Singapore
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore